CLINICAL TRIAL: NCT06016959
Title: Specialist Dietetic Intervention in Malnourished Patients with Fibrotic ILD: a Randomised Controlled Pilot Trial
Acronym: DT-ILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 327224
Record Dates: First submitted 2023-05-07; First posted 2023-08-30 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2023-10

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualised dietetic advice (Experimental): Participants will receive 5 sessions receiving individualised nutritional counselling advice from a registered dietitian.
  Interventions: Other: Dietetic intervention
- Diet sheet (Placebo Comparator): Participants will receive a diet sheet around poor appetite.
  Interventions: Other: Diet sheet (placebo)

INTERVENTIONS:
Other: Dietetic intervention — Dietetic intervention involves individualised and tailored dietary advice to patients struggling with their nutrition. This includes optimising energy and protein intake to improve malnutrition & also giving dietary advice to support with nutrition impact symptoms e.g. bloating.
  Arms: Individualised dietetic advice
Other: Diet sheet (placebo) — Patients randomised into the group receiving a diet sheet will be sent out Royal Brompton & Harefield Hospital's Poor Appetite diet booklet which involves general strategies to improve nutritional status (energy and protein)
  Arms: Diet sheet

SUMMARY:
Malnutrition occurs when the body receives too few nutrients, resulting in health problems such as weight loss. The consequences of malnutrition are worrying as they include lung failure, infection, and pressure ulcers.

Interstitial Lung Disease (ILD) is a term used for a group of diseases which can cause scarring of the lungs. Having ILD can cause malnutrition due to the lungs working hard and burning off energy. Additionally, medications called anti-fibrotic agents are used to slow disease progression. However, side effects include poor appetite, diarrhoea, nausea, vomiting and weight loss which can result in malnutrition.

Malnutrition occurs in ILD in approximately half of patients. This is important because the main signs of malnutrition such as weight loss and a low Body Mass Index (BMI), which takes into consideration your weight against your height, are linked with worse outcomes in ILD. Malnutrition in ILD can also reduce eligibility for lung transplant and can impact tolerability of anti-fibrotic agents. Research into treatment of malnutrition in ILD is limited.

Dietitians play a key role in diagnosis and treatment of malnutrition. This is because dietary counselling by a dietitian has been shown to increase quality of life and intake of energy in other chronic diseases. There are currently no studies documenting the benefits of dietetic intervention in patients with ILD.

We propose to undertake the first feasibility study in this area. A feasibility study is a first step trial which investigates whether a study can & should be done. The main aims of this study are:

1. How easy it is to recruit ILD patients to see a dietitian
2. Whether patients will attend dietetic appointments
3. Whether food/nutrient intake is increased following dietetic intervention
4. How acceptable is dietetic intervention to ILD patients As well as these main aims, this study will also provide initial information about whether dietetic intervention stabilises weight, BMI & quality of life.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 20kg/m2, or if aged >75, BMI ≤ 21 (Righini et al., 2013)
* Over the past 12 months, unintentional weight loss ≥ 5% of body weight, regardless of baseline BMI or weight loss >2 kg if BMI is normal.

Exclusion Criteria:

* Co-morbidities currently requiring a specialised diet (including enteral feeding)
* End of life care (estimated less than 6 weeks left to live)
* Expected introduction of anti-fibrotic or immunosuppressive treatment or introduction/increase corticosteroid dose during trial period
* Pregnancy
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 8 months
  Number individuals recruited/Number individuals contacted
Completion rate | 3 months
  Number individuals completing study/Number individuals randomised
Compliance | Defined by increased energy & protein intake versus run-in (three-day diet-diaries).
  3 months

SECONDARY OUTCOMES:
Nutritional status (Malnutrition) | 3 months
  PG-Subjective Global Assessment (SGA) which is a nutrition assessment tool using clinical parameters including weight loss, GI symptoms & functional capacity to diagnose malnutrition (Bauer et al., 2011).
Nutritional status (gastrointestinal related symptoms) | 3 months
  Gastrointestinal symptoms will be measured via the Gastrointestinal Symptom Rating Scale (GSRS) to further understand severity and impact of gastrointestinal related symptoms. (Svedlund et al., 1988)
Anthropometrics (weight) | 3 months
  Weight (kg) will be measured by VitaFit™ FCC/CE certified digital weighing scales provided during the first appointment or delivered at home, measured to an accuracy of 0.05kg. Dietitian led support for their use will be available.
Anthropometrics (height) | 3 months
  Height (m) will be derived from the most recent lung function reports.
Anthropometrics (Body Mass Index) | 3 months
  With the anthropometrics measured weight (kg) and height (m), this will be used to calculate Body Mass Index (BMI (kg/m2)).
Handgrip strength | 3 months
  Optimum nutrition can support maintenance of muscle to support activities of daily living. A CAMRY™ digital hand dynamometer will be delivered at home. HGS (kg) measures maximum voluntary muscle strength by squeezing the dynamometer providing a grip measurement accurate to 0.1kg.
Quality of Life (QoL) | 3 months
  Improved nutrition status may positively impact QoL. The King's Brief Interstitial Lung Disease Questionnaire (K-BILD), a 15-widely validated ILD-specific QoL questionnaire, will be used.
Energy and Protein intake | 3 months
  Participants will undertake a three-day diet diary at baseline and at 3 months to measure intake of macro and micronutrients will be calculated by using the software NutriticsTM, including daily total energy and protein intake as well as other nutrients, if necessary.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahai R, Castelli G, Danzo F, Ferreira L, Srirangan A, Morviducci M, Mirabelli FM, Kaenmuang P, Roberts C, Bax S, Hewitt RJ, Kokosi M, Chua F, Kouranos V, Molyneaux PL, George PM, Jenkins RG, Banya W, Stock CJW, Jones S, Korff G, Duncan A, Wells AU, Sestini P, Renzoni EA. Specialist Dietary Intervention in Patients With Fibrotic Interstitial Lung Disease Experiencing Unintentional Weight Loss: A Pilot Randomized Controlled Trial. Chest. 2025 Sep 25:S0012-3692(25)05388-7. doi: 10.1016/j.chest.2025.09.021. Online ahead of print. PMID 41015200